CLINICAL TRIAL: NCT00695656
Title: Profile of Hypertensive Patients Seen in General Practitioner Consultation
Brief Title: National Survey on Hypertension in General Practitioner (GP) Consultation
Acronym: Prophyl GP
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Alain Castaigne, Medical Director, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CFR-DUM-2007/7
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Hypertension
Keywords: Hypertension; general practitioner consultation; Patients with hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
To evaluate (with sufficient accuracy) the profile(demographic and clinical characteristics, health care management) of hypertensive patients seen in general practitioner consultation.

ELIGIBILITY:
Inclusion Criteria:

* male or female > or = 18 years old
* Known hypertension
* agree to take part in this study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First three consecutive patients with hypertension seen by general practitioner
Sampling Method: Probability Sample
Enrollment: 2853 (Actual)
Dates: Start 2008-04; Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Demographic, clinical and health care characteristics | Once

CONTACTS AND LOCATIONS:
Overall Officials: Castaigne, Medical Director, Study Director — AstraZeneca
Locations (1373):
- France (1373):
  - Research Site, Ablon-sur-Seine
  - Research Site, Agen
  - Research Site, Agneaux
  - Research Site, Agon-Coutainville
  - Research Site, Ahun
  - Research Site, Aiffres
  - Research Site, Aigueperse
  - Research Site, Aimargues
  - Research Site, Aire-sur-l'Adour
  - Research Site, Aire-sur-la-Lys
  - Research Site, Aix-en-Provence
  - Research Site, Aix-les-Bains
  - Research Site, Aixe-sur-Vienne
  - Research Site, Ajaccio
  - Research Site, Albert
  - Research Site, Alençon
  - Research Site, Alès
  - Research Site, Allaire
  - Research Site, Allouagne
  - Research Site, Althen-des-Paluds
  - Research Site, Amagne
  - Research Site, Ambert
  - Research Site, Ambès
  - Research Site, Ambierle
  - Research Site, Ambleteuse
  - Research Site, Amboise
  - Research Site, Amiens
  - Research Site, Amilly
  - Research Site, Amou
  - Research Site, Amphion-les-Bains
  - Research Site, Andeville
  - Research Site, Andres
  - Research Site, Anduze
  - Research Site, Angervilliers
  - Research Site, Angoulême
  - Research Site, Annecy-le-Vieux
  - Research Site, Annezin
  - Research Site, Annonay
  - Research Site, Ansauvillers
  - Research Site, Anse
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Ardres
  - Research Site, Argelès-Gazost
  - Research Site, Argenteuil
  - Research Site, Arles
  - Research Site, Arnage
  - Research Site, Arnèke
  - Research Site, Aron
  - Research Site, Arpajon
  - Research Site, Arras
  - Research Site, Arsac
  - Research Site, Artannes-sur-Indre
  - Research Site, Artix
  - Research Site, Arzacq-Arraziguet
  - Research Site, Aslonnes
  - Research Site, Athies
  - Research Site, Athis-Mons
  - Research Site, Aubagne
  - Research Site, Aubenas
  - Research Site, Aubervilliers
  - Research Site, Aubigny
  - Research Site, Aubin
  - Research Site, Auby
  - Research Site, Aucamville
  - Research Site, Auch
  - Research Site, Auchel
  - Research Site, Audincourt
  - Research Site, Audruicq
  - Research Site, Audun-le-Tiche
  - Research Site, Auffay
  - Research Site, Aulnat
  - Research Site, Aulnay-sous-Bois
  - Research Site, Aulnoy-lez-Valenciennes
  - Research Site, Aulnoye-Aymeries
  - Research Site, Aumont-Aubrac
  - Research Site, Auneau
  - Research Site, Auray
  - Research Site, Aussillon
  - Research Site, Auvers-sur-Oise
  - Research Site, Auxerre
  - Research Site, Auxi-le-Château
  - Research Site, Availles-Limouzine
  - Research Site, Avallon
  - Research Site, Avenay-Val-d'Or
  - Research Site, Avesnes-le-Sec
  - Research Site, Avesnes-les-Aubert
  - Research Site, Avion
  - Research Site, Avon
  - Research Site, Avrillé
  - Research Site, Bagnères-de-Bigorre
  - Research Site, Bagnols-sur-Cèze
  - Research Site, Baignes STE Radegonde
  - Research Site, Baincthun
  - Research Site, Bains
  - Research Site, Balma
  - Research Site, Bandol
  - Research Site, Barbezieux-Saint-Hilaire
  - Research Site, Barjols
  - Research Site, Barneville-Carteret
  - Research Site, Basse Pointe
  - Research Site, Bassens
  - Research Site, Bassillac
  - Research Site, Bastia
  - Research Site, Batz-sur-Mer
  - Research Site, Baume-les-Dames
  - Research Site, Bauvin
  - Research Site, Bayeux
  - Research Site, Beaulieu-sous-la-Roche
  - Research Site, Beaumes-de-Venise
  - Research Site, Beaumont-en-Véron
  - Research Site, Beaumont-sur-Oise
  - Research Site, Beaurepaire
  - Research Site, Beaurieux
  - Research Site, Beautor
  - Research Site, Beauvais
  - Research Site, Beauvoir-sur-Niort
  - Research Site, Behren-lès-Forbach
  - Research Site, Belfort
  - Research Site, Bellac
  - Research Site, Benfeld
  - Research Site, Bennecourt
  - Research Site, Bergerac
  - Research Site, Berlaimont
  - Research Site, Bernay
  - Research Site, Berrwiller
  - Research Site, Bertrichamps
  - Research Site, Bessières
  - Research Site, Bettancourt-la-Ferrée
  - Research Site, Betton
  - Research Site, Bezouce
  - Research Site, Bégard
  - Research Site, Bétaille
  - Research Site, Béthune
  - Research Site, Bézenet
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Bidart
  - Research Site, Biganos
  - Research Site, Binic
  - Research Site, Bischwiller
  - Research Site, Blagnac
  - Research Site, Blangy-sur-Bresle
  - Research Site, Blanzy
  - Research Site, Blois
  - Research Site, Bogny-sur-Meuse
  - Research Site, Bois-Guillaume
  - Research Site, Boissy-Saint-Léger
  - Research Site, Bolbec
  - Research Site, Bondues
  - Research Site, Bonneuil-sur-Marne
  - Research Site, Bonnières-sur-Seine
  - Research Site, Bonny-sur-Loire
  - Research Site, Bordeaux
  - Research Site, Borgo
  - Research Site, Bormes-les-Mimosas
  - Research Site, Bosc-le-Hard
  - Research Site, Bouafle
  - Research Site, Bouchet
  - Research Site, Boulange
  - Research Site, Bouliac
  - Research Site, Boulogne-sur-Mer
  - Research Site, Bourbourg
  - Research Site, Bourg de Joué-sur-Erdre
  - Research Site, Bourg-en-Bresse
  - Research Site, Bourg-la-Reine
  - Research Site, Bourges
  - Research Site, Bourré
  - Research Site, Bouvron
  - Research Site, Bozouls
  - Research Site, Braine
  - Research Site, Branne
  - Research Site, Brantôme
  - Research Site, Brax
  - Research Site, Brens
  - Research Site, Bresles
  - Research Site, Brest
  - Research Site, Breteuil
  - Research Site, Bretteville-sur-Odon
  - Research Site, Breuil-le-Sec
  - Research Site, Bréhal
  - Research Site, Briançon
  - Research Site, Brignon
  - Research Site, Brignoud
  - Research Site, Brioude
  - Research Site, Brocas
  - Research Site, Broût-Vernet
  - Research Site, Bruère-Allichamps
  - Research Site, Bruges
  - Research Site, Brumath
  - Research Site, Brunehamel
  - Research Site, Brunoy
  - Research Site, Brunstatt
  - Research Site, Bucquoy
  - Research Site, Bully-les-Mines
  - Research Site, Buxerolles
  - Research Site, Buxières-les-Mines
  - Research Site, Cadenet
  - Research Site, Caen
  - Research Site, Cagnes-sur-Mer
  - Research Site, Cailly
  - Research Site, Camblanes
  - Research Site, Cambo-les-Bains
  - Research Site, Cambrai
  - Research Site, Cambrin
  - Research Site, Canet-Plage
  - Research Site, Canéjan
  - Research Site, Cannes
  - Research Site, Canohès
  - Research Site, Capbreton
  - Research Site, Capdenac-Gare
  - Research Site, Carbon-Blanc
  - Research Site, Carcassonne
  - Research Site, Carcès
  - Research Site, Carentan
  - Research Site, Carhaix-Plouguer
  - Research Site, Caro
  - Research Site, Carpentras
  - Research Site, Carpiquet
  - Research Site, Carrières-sur-Seine
  - Research Site, Carros
  - Research Site, Carrouges
  - Research Site, Carry-le-Rouet
  - Research Site, Carvin
  - Research Site, CASE Pilote
  - Research Site, Castanet-Tolosan
  - Research Site, Castelnaudary
  - Research Site, Castelsarrasin
  - Research Site, Castillon-la-Bataille
  - Research Site, Castres
  - Research Site, Caudiès-de-Fenouillèdes
  - Research Site, Caylus
  - Research Site, Cayriech
  - Research Site, Celles-sur-Durolle
  - Research Site, Celles-sur-Plaine
  - Research Site, Cepoy
  - Research Site, Cergy
  - Research Site, Ceyreste
  - Research Site, Chaillevette
  - Research Site, Chalais
  - Research Site, Chaleins
  - Research Site, Challain-la-Potherie
  - Research Site, Chalon-sur-Saône
  - Research Site, Chambéry
  - Research Site, Chambray-lès-Tours
  - Research Site, Champagné
  - Research Site, Champcueil
  - Research Site, Champigneulles
  - Research Site, Champigné
  - Research Site, Champvans
  - Research Site, Chancelade
  - Research Site, Changé
  - Research Site, Chantilly
  - Research Site, Chantonnay
  - Research Site, Chapelle Saint Martin Plaine
  - Research Site, Chaponost
  - Research Site, Charleville-Mézières
  - Research Site, Charmes
  - Research Site, Chartres
  - Research Site, Chateauneuf ILLE Vilaine
  - Research Site, Chauffailles
  - Research Site, Chaumergy
  - Research Site, Chaumont
  - Research Site, Chauvigny
  - Research Site, Chavanay
  - Research Site, Chazay-d'Azergues
  - Research Site, Châbons
  - Research Site, Château-Chinon(Ville)
  - Research Site, Château-Gontier
  - Research Site, Château-Landon
  - Research Site, Château-Porcien
  - Research Site, Château-Renard
  - Research Site, Château-Thierry
  - Research Site, Châteaubriant
  - Research Site, Châteauneuf-du-Pape
  - Research Site, Châteauneuf-en-Thymerais
  - Research Site, Châteauneuf-sur-Cher
  - Research Site, Châteauroux
  - Research Site, Châtelaudren
  - Research Site, Châtellerault
  - Research Site, Châtenay-Malabry
  - Research Site, Châtillon-Coligny
  - Research Site, Châtillon-sur-Colmont
  - Research Site, Cheminot
  - Research Site, Cherves-Richemont
  - Research Site, Chevilly
  - Research Site, Chéreng
  - Research Site, Choisy-le-Roi
  - Research Site, Cholet
  - Research Site, Ciry-le-Noble
  - Research Site, Civray
  - Research Site, Clamart
  - Research Site, Clary
  - Research Site, Clermont-Ferrand
  - Research Site, Cléon-d'Andran
  - Research Site, Clichy
  - Research Site, Clichy-sous-Bois
  - Research Site, Cluses
  - Research Site, Collioure
  - Research Site, Colmar
  - Research Site, Colomiers
  - Research Site, Combs-la-Ville
  - Research Site, Comines
  - Research Site, Commelle
  - Research Site, Concarneau
  - Research Site, Condé-en-Brie
  - Research Site, Confolens
  - Research Site, Contamine-sur-Arve
  - Research Site, Contres
  - Research Site, Coquelles
  - Research Site, Corbehem
  - Research Site, Corbeil-Essonnes
  - Research Site, Corbeny
  - Research Site, Cormoranche-sur-Saône
  - Research Site, Corrèze
  - Research Site, Corseul
  - Research Site, Cosne-Cours-sur-Loire
  - Research Site, Coubon
  - Research Site, Couëron
  - Research Site, Couhé
  - Research Site, Coulommiers
  - Research Site, Courbevoie
  - Research Site, Cournon-d'Auvergne
  - Research Site, Courpière
  - Research Site, Coutouvre
  - Research Site, Coutras
  - Research Site, Couzeix
  - Research Site, Coye-la-Forêt
  - Research Site, Crèvecœur-le-Grand
  - Research Site, Crécy-en-Ponthieu
  - Research Site, Créteil
  - Research Site, Criquetot-l'Esneval
  - Research Site, Croix
  - Research Site, Cros-de-Cagnes
  - Research Site, Crosne
  - Research Site, Cubjac
  - Research Site, Cublac
  - Research Site, Cugand
  - Research Site, Cugnaux
  - Research Site, Cuincy
  - Research Site, Cysoing
  - Research Site, Dainville
  - Research Site, Dambach-la-Ville
  - Research Site, Danjoutin
  - Research Site, Dannemarie
  - Research Site, Dax
  - Research Site, Deauville
  - Research Site, Decazeville
  - Research Site, Denain
  - Research Site, Deyvillers
  - Research Site, Déville-lès-Rouen
  - Research Site, Diarville
  - Research Site, Dieppe
  - Research Site, Dieulefit
  - Research Site, Dieuze
  - Research Site, Digoin
  - Research Site, Dinard
  - Research Site, Divion
  - Research Site, Dolus-d'Oléron
  - Research Site, Domfront
  - Research Site, Domont
  - Research Site, Donzy
  - Research Site, Douai
  - Research Site, Douarnenez
  - Research Site, Doucier
  - Research Site, Doué-la-Fontaine
  - Research Site, Douvaine
  - Research Site, Draguignan
  - Research Site, Drancy
  - Research Site, Drumettaz
  - Research Site, Drusenheim
  - Research Site, Ducos
  - Research Site, Dunières
  - Research Site, Durban-Corbières
  - Research Site, Eaubonne
  - Research Site, Elliant
  - Research Site, Entraygues-sur-Truyère
  - Research Site, Entrevaux
  - Research Site, Ermont
  - Research Site, Escaudain
  - Research Site, Espalion
  - Research Site, Estagel
  - Research Site, Estivareilles
  - Research Site, Eu
  - Research Site, Eymoutiers
  - Research Site, Échirolles
  - Research Site, Écommoy
  - Research Site, Écouché
  - Research Site, Écouflant
  - Research Site, Écully
  - Research Site, Égletons
  - Research Site, Épernon
  - Research Site, Épinac
  - Research Site, Épinal
  - Research Site, Épinay-sur-Orge
  - Research Site, Épinay-sur-Seine
  - Research Site, Équeurdreville-Hainneville
  - Research Site, Étalondes
  - Research Site, Étampes
  - Research Site, Étaples
  - Research Site, Étival-Clairefontaine
  - Research Site, Évaux-les-Bains
  - Research Site, Évron
  - Research Site, Ézy-sur-Eure
  - Research Site, Faverges
  - Research Site, Fayence
  - Research Site, Fegersheim
  - Research Site, Felletin
  - Research Site, Fenouillet
  - Research Site, Ferrière-la-Grande
  - Research Site, Feurs
  - Research Site, Fécamp
  - Research Site, Firmi
  - Research Site, Firminy
  - Research Site, Flayosc
  - Research Site, Flers
  - Research Site, Fleury
  - Research Site, Fleury-sur-Orne
  - Research Site, Flixecourt
  - Research Site, Floing
  - Research Site, Florange
  - Research Site, Florensac
  - Research Site, Fontaine-lès-Dijon
  - Research Site, Fontenay-en-Parisis
  - Research Site, Fontenay-sous-Bois
  - Research Site, FORT de France Cedex
  - Research Site, FORT de France
  - Research Site, Fos-sur-Mer
  - Research Site, Fosses
  - Research Site, Fougères
  - Research Site, Fourchambault
  - Research Site, Fourmies
  - Research Site, Foussais-Payré
  - Research Site, Franconville
  - Research Site, Frangy
  - Research Site, Frasne
  - Research Site, Fresnes-sur-Escaut
  - Research Site, Fréjus
  - Research Site, Fréland
  - Research Site, Froideconche
  - Research Site, Fromentine
  - Research Site, Fumay
  - Research Site, Fussy
  - Research Site, Gabian
  - Research Site, Gacé
  - Research Site, Gaillac
  - Research Site, Gaillon
  - Research Site, Gallardon
  - Research Site, Ganges
  - Research Site, Gardonne
  - Research Site, Garéoult
  - Research Site, Gargas
  - Research Site, Garges-lès-Gonesse
  - Research Site, Gauriac
  - Research Site, Gelles
  - Research Site, Gelos
  - Research Site, Genlis
  - Research Site, Gennevilliers
  - Research Site, Gerzat
  - Research Site, Gex
  - Research Site, Gien
  - Research Site, Gignac-la-Nerthe
  - Research Site, Giraumont
  - Research Site, Gironde-sur-Dropt
  - Research Site, Givrand
  - Research Site, Goderville
  - Research Site, Golbey
  - Research Site, Gonneville-la-Mallet
  - Research Site, Gontaud-de-Nogaret
  - Research Site, Goussainville
  - Research Site, Gouvieux
  - Research Site, Grand-Champ
  - Research Site, Grandvillars
  - Research Site, Granges-sur-Vologne
  - Research Site, Graulhet
  - Research Site, Gravelines
  - Research Site, Gray-la-Ville
  - Research Site, Grayan
  - Research Site, Grenade
  - Research Site, Grenoble
  - Research Site, Gréasque
  - Research Site, Gries
  - Research Site, Griesheim-près-Molsheim
  - Research Site, Grignols
  - Research Site, Grisolles
  - Research Site, Groisy
  - Research Site, Grosbliederstroff
  - Research Site, Groslay
  - Research Site, Guebwiller
  - Research Site, Guerlesquin
  - Research Site, Guérande
  - Research Site, Guéret
  - Research Site, Guignicourt
  - Research Site, Guipavas
  - Research Site, Guînes
  - Research Site, Gujan-Mestras
  - Research Site, Gurmençon
  - Research Site, Gy
  - Research Site, Hagetmau
  - Research Site, Hagondange
  - Research Site, Haguenau
  - Research Site, Halluin
  - Research Site, Ham
  - Research Site, Ham-en-Artois
  - Research Site, Hangenbieten
  - Research Site, Harnes
  - Research Site, Haroué
  - Research Site, Hasparren
  - Research Site, Hatten
  - Research Site, Hattenville
  - Research Site, Hauteville-Lompnes
  - Research Site, Hautmont
  - Research Site, Hem
  - Research Site, Herbault
  - Research Site, Herbignac
  - Research Site, Hettange-Grande
  - Research Site, Hégenheim
  - Research Site, Hénin-Beaumont
  - Research Site, Hochstatt
  - Research Site, Holtzheim
  - Research Site, Honfleur
  - Research Site, Houdain
  - Research Site, Houplin-Ancoisne
  - Research Site, Hundling
  - Research Site, Hyères
  - Research Site, Ibos
  - Research Site, Illiers-Combray
  - Research Site, Irigny
  - Research Site, Isle
  - Research Site, Issy-les-Moulineaux
  - Research Site, Istres
  - Research Site, Ivry-sur-Seine
  - Research Site, Janzé
  - Research Site, Jardin
  - Research Site, Jarny
  - Research Site, Jarville-la-Malgrange
  - Research Site, Jaunay-Clan
  - Research Site, Joyeuse
  - Research Site, Juniville
  - Research Site, Kingersheim
  - Research Site, L'Étrat
  - Research Site, L'Isle-Adam
  - Research Site, L'Isle-Jourdain
  - Research Site, La Baule-Escoublac
  - Research Site, La Bouilladisse
  - Research Site, La Bruffière
  - Research Site, La Canourgue
  - Research Site, La Chambre
  - Research Site, La Chapelle-des-Fougeretz
  - Research Site, La Ciotat
  - Research Site, La Claquette
  - Research Site, La Clayette
  - Research Site, La Courneuve
  - Research Site, La Crau
  - Research Site, La Fare-les-Oliviers
  - Research Site, La Ferté-Bernard
  - Research Site, La Ferté-Gaucher
  - Research Site, La Ferté-sous-Jouarre
  - Research Site, La Flotte
  - Research Site, La Fouillade
  - Research Site, La Francheville
  - Research Site, La Frenaye
  - Research Site, La Fresnaye-sur-Chédouet
  - Research Site, La Frette
  - Research Site, La Garde
  - Research Site, La Garnache
  - Research Site, La Génétouze
  - Research Site, La Grand-Combe
  - Research Site, La Grande-Motte
  - Research Site, La Haye-du-Puits
  - Research Site, La Haye-Malherbe
  - Research Site, La Haye-Pesnel
  - Research Site, La Londe-les-Maures
  - Research Site, La Loupe
  - Research Site, La Mailleraye-sur-Seine
  - Research Site, La Membrolle-sur-Choisille
  - Research Site, La Mothe-Saint-Héray
  - Research Site, La Mulatière
  - Research Site, La Neuville-Roy
  - Research Site, La Pommeraye
  - Research Site, La Réole
  - Research Site, La Riche
  - Research Site, La Roche-sur-Yon
  - Research Site, La Rochefoucauld
  - Research Site, La Rochelle
  - Research Site, La Roquebrussanne
  - Research Site, La Seyne-sur-Mer
  - Research Site, La Source
  - Research Site, La Souterraine
  - Research Site, La Teste-de-Buch
  - Research Site, La Trinité
  - Research Site, La Ville-Dieu-du-Temple
  - Research Site, Labarthe-Rivière
  - Research Site, Labastide-Murat
  - Research Site, Labastide-Saint-Pierre
  - Research Site, Lablachère
  - Research Site, Labouheyre
  - Research Site, Lacapelle-Biron
  - Research Site, Lacaune
  - Research Site, Lacrouzette
  - Research Site, Laillé
  - Research Site, Laissac
  - Research Site, Lamagistère
  - Research Site, Lambersart
  - Research Site, Lançon-Provence
  - Research Site, Landas
  - Research Site, Landerneau
  - Research Site, Landes
  - Research Site, Landouge
  - Research Site, Landrecies
  - Research Site, Langres
  - Research Site, Lannion
  - Research Site, Lannoy
  - Research Site, Lanvéoc
  - Research Site, Lanvollon
  - Research Site, Laon
  - Research Site, Lapugnoy
  - Research Site, Laure
  - Research Site, Laxou
  - Research Site, Lay-Saint-Christophe
  - Research Site, Le Barp
  - Research Site, Le Blanc-Mesnil
  - Research Site, Le Bois-dOingt
  - Research Site, Le Boulou
  - Research Site, Le Bouscat
  - Research Site, Le Bugue
  - Research Site, Le Cannet
  - Research Site, Le Chambon-Feugerolles
  - Research Site, Le Châtelet-en-Brie
  - Research Site, Le Clion-sur-Mer
  - Research Site, LE Diamant
  - Research Site, Le Donjon
  - Research Site, Le Dorat
  - Research Site, Le Fenouiller
  - Research Site, Le Frasnois
  - Research Site, LE Golfe JUAN
  - Research Site, Le Grand-Lemps
  - Research Site, Le Grand-Quevilly
  - Research Site, Le Havre
  - Research Site, LE Lamentin
  - Research Site, Le Lardin-Saint-Lazare
  - Research Site, Le Lavandou
  - Research Site, LE Lorrain
  - Research Site, Le Luc
  - Research Site, Le Lude
  - Research Site, Le Mans
  - Research Site, LE Marin
  - Research Site, Le May-sur-Èvre
  - Research Site, Le Mayet-de-Montagne
  - Research Site, Le Monastier-sur-Gazeille
  - Research Site, LE Morne Rouge
  - Research Site, Le Neubourg
  - Research Site, Le Perray-en-Yvelines
  - Research Site, Le Perreux-sur-Marne
  - Research Site, Le Péage-de-Roussillon
  - Research Site, Le Plessis-Trévise
  - Research Site, Le Pont-de-Beauvoisin
  - Research Site, Le Pouliguen
  - Research Site, Le Rove
  - Research Site, Le Russey
  - Research Site, Le Sap
  - Research Site, Le Soler
  - Research Site, Le Taillan-Médoc
  - Research Site, Le Teil
  - Research Site, Le Thor
  - Research Site, Le Touquet-Paris-Plage
  - Research Site, Le Touvet
  - Research Site, Le Veurdre
  - Research Site, Lectoure
  - Research Site, Leers
  - Research Site, Leforest
  - Research Site, Lens
  - Research Site, Les Ancizes
  - Research Site, Les Avenières
  - Research Site, Les Forges
  - Research Site, Les Hautes-Rivières
  - Research Site, Les Montils
  - Research Site, Les Mureaux
  - Research Site, Les Pennes-Mirabeau
  - Research Site, Les Pieux
  - Research Site, Les Ponts-de-Cé
  - Research Site, Les Sables-d'Olonne
  - Research Site, Les Touches
  - Research Site, LES Trois Ilets
  - Research Site, Lesparre-Médoc
  - Research Site, Levier
  - Research Site, Levroux
  - Research Site, Lexy
  - Research Site, Lezoux
  - Research Site, Lédignan
  - Research Site, Léry
  - Research Site, Lézardrieux
  - Research Site, Lézignan-Corbières
  - Research Site, Liancourt
  - Research Site, Libercourt
  - Research Site, Libourne
  - Research Site, LIEU DIT Carnon Plage
  - Research Site, Liévin
  - Research Site, Liffol-le-Grand
  - Research Site, Lignan-sur-Orb
  - Research Site, Lillebonne
  - Research Site, Limeil-Brévannes
  - Research Site, Limoges
  - Research Site, Limogne-en-Quercy
  - Research Site, Limoux
  - Research Site, Lingolsheim
  - Research Site, Linselles
  - Research Site, Lisieux
  - Research Site, Livarot
  - Research Site, Loches
  - Research Site, Locmiquélic
  - Research Site, Locon
  - Research Site, Lodève
  - Research Site, Longueau
  - Research Site, Loos-en-Gohelle
  - Research Site, Lorient
  - Research Site, Loudes
  - Research Site, Loué
  - Research Site, Loulay
  - Research Site, Lourdes
  - Research Site, Loures-Barousse
  - Research Site, Loyettes
  - Research Site, Luant
  - Research Site, Lunéville
  - Research Site, Lurcy-Lévis
  - Research Site, Lusignan
  - Research Site, Lussac-les-Châteaux
  - Research Site, Luxé
  - Research Site, Lyon
  - Research Site, Lys-lez-Lannoy
  - Research Site, Mably
  - Research Site, Magnac-Bourg
  - Research Site, Magné
  - Research Site, Maintenon
  - Research Site, Mainvilliers
  - Research Site, Maizières-lès-Metz
  - Research Site, Maîche
  - Research Site, Malissard
  - Research Site, Mandres-les-Roses
  - Research Site, Manduel
  - Research Site, Mansle
  - Research Site, Mantes-la-Jolie
  - Research Site, Marans
  - Research Site, Maraussan
  - Research Site, Marciac
  - Research Site, Marcorignan
  - Research Site, Marcq-en-Barœul
  - Research Site, Marignane
  - Research Site, Marignier
  - Research Site, Marle
  - Research Site, Marlenheim
  - Research Site, Marmande
  - Research Site, Maromme
  - Research Site, Marquion
  - Research Site, Mars-la-Tour
  - Research Site, Marsannay-la-Côte
  - Research Site, Marseillan Plage
  - Research Site, Marseille
  - Research Site, Marthon
  - Research Site, Martigues
  - Research Site, Marvejols
  - Research Site, Mas-Grenier
  - Research Site, Masseret
  - Research Site, Matignon
  - Research Site, Maubourguet
  - Research Site, Mauguio
  - Research Site, Mauléon-Licharre
  - Research Site, Maury
  - Research Site, Mauvezin
  - Research Site, Maxéville
  - Research Site, Mazamet
  - Research Site, Mazan
  - Research Site, Mâcon
  - Research Site, Meaux
  - Research Site, Melgven
  - Research Site, Mennevret
  - Research Site, Merkwiller-Pechelbronn
  - Research Site, Merlines
  - Research Site, Merry-la-Vallée
  - Research Site, Mers-les-Bains
  - Research Site, Mertzwiller
  - Research Site, Mervent
  - Research Site, Merville
  - Research Site, Mesvres
  - Research Site, Metz
  - Research Site, Metzervisse
  - Research Site, Meursac
  - Research Site, Meymac
  - Research Site, Mezel
  - Research Site, Mezzavia
  - Research Site, Mérignac
  - Research Site, Mézidon-Canon
  - Research Site, Mézilles
  - Research Site, Millau
  - Research Site, Mimizan
  - Research Site, Miramas
  - Research Site, Miramont-de-Guyenne
  - Research Site, Mirande
  - Research Site, Missillac
  - Research Site, Mittersheim
  - Research Site, Molières
  - Research Site, Moncé-en-Belin
  - Research Site, Moncrabeau
  - Research Site, Mondelange
  - Research Site, Mons
  - Research Site, Mons-en-Laonnois
  - Research Site, Mons-en-Pévèle
  - Research Site, Mont-de-Marsan
  - Research Site, Mont-Saint-Martin
  - Research Site, Montady
  - Research Site, Montaigut
  - Research Site, Montauban
  - Research Site, Montauroux
  - Research Site, Montbazens
  - Research Site, Montbazin
  - Research Site, Montbéliard
  - Research Site, Montbrison
  - Research Site, Montceau-les-Mines
  - Research Site, Montdidier
  - Research Site, Montélimar
  - Research Site, Montfavet
  - Research Site, Montfort-en-Chalosse
  - Research Site, Montfort-sur-Risle
  - Research Site, Montguyon
  - Research Site, Monthermé
  - Research Site, Montigny-en-Ostrevent
  - Research Site, Montigny-le-Roi
  - Research Site, Montigny-lès-Cormeilles
  - Research Site, Montigny-lès-Metz
  - Research Site, Montlouis-sur-Loire
  - Research Site, Montluçon
  - Research Site, Montmirail
  - Research Site, Montmorillon
  - Research Site, Montmorot
  - Research Site, Montpellier
  - Research Site, Montrabé
  - Research Site, Montret
  - Research Site, Montreuil
  - Research Site, Monts-sur-Guesnes
  - Research Site, Morangis
  - Research Site, Morlaix
  - Research Site, Mortagne-sur-Gironde
  - Research Site, Mortain
  - Research Site, Moulins
  - Research Site, Moussac
  - Research Site, Moutiers-les-Mauxfaits
  - Research Site, Mouvaux
  - Research Site, Mulhouse
  - Research Site, Nançay
  - Research Site, Nans-les-Pins
  - Research Site, Nanterre
  - Research Site, Nantes
  - Research Site, Nanteuil-en-Vallée
  - Research Site, Narbonne
  - Research Site, Naucelle
  - Research Site, Nay
  - Research Site, Nemours
  - Research Site, Neuf-Mesnil
  - Research Site, Neufchef
  - Research Site, Neuilly-sur-Seine
  - Research Site, Neuville-en-Ferrain
  - Research Site, Neuville-les-Dames
  - Research Site, Neuville-Saint-Rémy
  - Research Site, Neuvillette
  - Research Site, Nevers
  - Research Site, Nexon
  - Research Site, Nègrepelisse
  - Research Site, Nérac
  - Research Site, Nice
  - Research Site, Niederbronn-les-Bains
  - Research Site, Nilvange
  - Research Site, Niort
  - Research Site, Noé
  - Research Site, Nogent-le-Phaye
  - Research Site, Noirmoutier-en-l'Île
  - Research Site, Noisy-le-Grand
  - Research Site, Nontron
  - Research Site, Nordausques
  - Research Site, Novéant-sur-Moselle
  - Research Site, Noyal-Pontivy
  - Research Site, Noyen-sur-Sarthe
  - Research Site, Noyers-Bocage
  - Research Site, Noyers-sur-Cher
  - Research Site, Nozay
  - Research Site, Oberhausbergen
  - Research Site, Ohlungen
  - Research Site, Oignies
  - Research Site, Oisemont
  - Research Site, Ollioules
  - Research Site, Orange
  - Research Site, Orbec
  - Research Site, Orcines
  - Research Site, Origny STE Benoite
  - Research Site, Orléans
  - Research Site, Orliénas
  - Research Site, Orly
  - Research Site, Ormesson-sur-Marne
  - Research Site, Orthez
  - Research Site, Oullins
  - Research Site, Oye-Plage
  - Research Site, Oyonnax
  - Research Site, Pagny-sur-Moselle
  - Research Site, Paimboeuf
  - Research Site, Paimpol
  - Research Site, Paimpont
  - Research Site, Pamproux
  - Research Site, Pantin
  - Research Site, Parempuyre
  - Research Site, Paris
  - Research Site, Pas-en-Artois
  - Research Site, Pau
  - Research Site, Pauillac
  - Research Site, Pavilly
  - Research Site, Pecquencourt
  - Research Site, Pellegrue
  - Research Site, Pennautier
  - Research Site, Pernes-les-Fontaines
  - Research Site, Perpignan
  - Research Site, Perriers-sur-Andelle
  - Research Site, Petit-Noir
  - Research Site, Peyriac-de-Mer
  - Research Site, Pénestin
  - Research Site, Périers
  - Research Site, Périgueux
  - Research Site, Pérols
  - Research Site, Phalsbourg
  - Research Site, Pibrac
  - Research Site, Pierrefitte-sur-Seine
  - Research Site, Pitgam
  - Research Site, Pithiviers
  - Research Site, Plabennec
  - Research Site, Plan-de-Cuques
  - Research Site, Plaudren
  - Research Site, Plauzat
  - Research Site, Plessala
  - Research Site, Pleumeur-Gautier
  - Research Site, Pleurtuit
  - Research Site, Ploeren
  - Research Site, Plouarzel
  - Research Site, Plouay
  - Research Site, Ploudaniel
  - Research Site, Plouha
  - Research Site, Plouigneau
  - Research Site, Plourivo
  - Research Site, Plouzané
  - Research Site, Plouzévédé
  - Research Site, Pluvigner
  - Research Site, Pocé-sur-Cisse
  - Research Site, Poissy
  - Research Site, Polliat
  - Research Site, Poncin
  - Research Site, Pont-Audemer
  - Research Site, Pont-à-Mousson
  - Research Site, Pont-d'Ouilly
  - Research Site, Pont-de-l'Arche
  - Research Site, Pont-de-Vaux
  - Research Site, Pont-de-Veyle
  - Research Site, Pont-Évêque
  - Research Site, Pont-l'Abbé-d'Arnoult
  - Research Site, Pont-l'Évêque
  - Research Site, Pont-Saint-Pierre
  - Research Site, Pont-sur-Sambre
  - Research Site, Pontcharra
  - Research Site, Pontcharra-sur-Turdine
  - Research Site, Pontchâteau
  - Research Site, Pontenx-les-Forges
  - Research Site, Pontgibaud
  - Research Site, Pontivy
  - Research Site, Pordic
  - Research Site, Pornic
  - Research Site, Pornichet
  - Research Site, Port Leucate
  - Research Site, Port-La Nouvelle
  - Research Site, Pougues-les-Eaux
  - Research Site, Pouillon
  - Research Site, Pouldreuzic
  - Research Site, Pouzay
  - Research Site, Prades
  - Research Site, Pradines
  - Research Site, Presles
  - Research Site, Pringy
  - Research Site, Privas
  - Research Site, Puget-sur-Argens
  - Research Site, Puget-Ville
  - Research Site, Puisserguier
  - Research Site, Putanges-Pont-Écrepin
  - Research Site, Querqueville
  - Research Site, Quiévy
  - Research Site, Quimper
  - Research Site, Quimperlé
  - Research Site, Quincy-sous-Sénart
  - Research Site, Quintin
  - Research Site, Raismes
  - Research Site, Rambervillers
  - Research Site, Ravières
  - Research Site, Redon
  - Research Site, Reims
  - Research Site, Remiremont
  - Research Site, Remy
  - Research Site, Renazé
  - Research Site, Rennes
  - Research Site, Revel
  - Research Site, Revin
  - Research Site, Riantec
  - Research Site, Richemont
  - Research Site, Riedisheim
  - Research Site, Rieupeyroux
  - Research Site, Riom
  - Research Site, Rioupéroux
  - Research Site, Ris-Orangis
  - Research Site, Rivehaute
  - Research Site, Riviere Pilote
  - Research Site, Rivière-sur-Tarn
  - Research Site, Roanne
  - Research Site, Robert VERT PRE
  - Research Site, Robion
  - Research Site, Rocbaron
  - Research Site, Roche-la-Molière
  - Research Site, Rodez
  - Research Site, Rognes
  - Research Site, Rohrbach-lès-Bitche
  - Research Site, Roisel
  - Research Site, Roissy-en-Brie
  - Research Site, Romainville
  - Research Site, Romans-sur-Isère
  - Research Site, Rombas
  - Research Site, Romorantin-Lanthenay
  - Research Site, Roncq
  - Research Site, Roquebrune-Cap-Martin
  - Research Site, Roquefort-la-Bédoule
  - Research Site, Roquefort-sur-Soulzon
  - Research Site, Rosières-en-Santerre
  - Research Site, Rosny-sur-Seine
  - Research Site, Roubaix
  - Research Site, Rouen
  - Research Site, Roullet-Saint-Estèphe
  - Research Site, Roumazières
  - Research Site, Rousson
  - Research Site, Roye
  - Research Site, Rozay-en-Brie
  - Research Site, Rozier-en-Donzy
  - Research Site, Rueil-Malmaison
  - Research Site, Rully
  - Research Site, Sabres
  - Research Site, Saint Georges Baillargeaux
  - Research Site, Saint Maximin LA STE Baume
  - Research Site, Saint-Affrique
  - Research Site, Saint-Alban-de-Montbel
  - Research Site, Saint-Amand-en-Puisaye
  - Research Site, Saint-Ambroix
  - Research Site, Saint-Amé
  - Research Site, Saint-André-de-Corcy
  - Research Site, Saint-André-de-Sangonis
  - Research Site, Saint-Anthème
  - Research Site, Saint-Aubin-de-Médoc
  - Research Site, Saint-Aubin-des-Châteaux
  - Research Site, Saint-Aubin-le-Cloud
  - Research Site, Saint-Aubin-sur-Mer
  - Research Site, Saint-Augustin
  - Research Site, Saint-Avertin
  - Research Site, Saint-Aygulf
  - Research Site, Saint-Barthélémy
  - Research Site, Saint-Beauzély
  - Research Site, Saint-Berthevin
  - Research Site, Saint-Bonnet-sur-Gironde
  - Research Site, Saint-Brevin-les-Pins
  - Research Site, Saint-Brice-Courcelles
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Caradec
  - Research Site, Saint-Chély-d'Apcher
  - Research Site, Saint-Ciers-sur-Gironde
  - Research Site, Saint-Claude
  - Research Site, Saint-Cloud
  - Research Site, Saint-Cyr-sur-Loire
  - Research Site, Saint-Cyr-sur-Mer
  - Research Site, Saint-Denis
  - Research Site, Saint-Denis-de-Jouhet
  - Research Site, Saint-Denis-lès-Bourg
  - Research Site, Saint-Dizier
  - Research Site, Saint-Doulchard
  - Research Site, Saint-Esprit
  - Research Site, Saint-Etienne
  - Research Site, Saint-Etienne-de-Tulmont
  - Research Site, Saint-Étienne-de-Montluc
  - Research Site, Saint-Fort-sur-Gironde
  - Research Site, Saint-Georges-de-Didonne
  - Research Site, Saint-Georges-la-Pouge
  - Research Site, Saint-Germain-du-Plain
  - Research Site, Saint-Germain-les-Belles
  - Research Site, Saint-Germain-lès-Corbeil
  - Research Site, Saint-Germainmont
  - Research Site, Saint-Gervais-d'Auvergne
  - Research Site, Saint-Guénolé
  - Research Site, Saint-Herblon
  - Research Site, Saint-Hilaire-de-Brethmas
  - Research Site, Saint-Hilaire-de-Riez
  - Research Site, Saint-Hippolyte-du-Fort
  - Research Site, Saint-Jacques-sur-Darnétal
  - Research Site, Saint-Jean-de-Luz
  - Research Site, Saint-Jean-de-Maurienne
  - Research Site, Saint-Jean-de-Sixt
  - Research Site, Saint-Jean-de-Védas
  - Research Site, Saint-Jean-en-Royans
  - Research Site, Saint-Joseph
  - Research Site, Saint-Julien-l'Ars
  - Research Site, Saint-Just-Chaleyssin
  - Research Site, Saint-Just-en-Chaussée
  - Research Site, Saint-Just-le-Martel
  - Research Site, Saint-Laurent-Blangy
  - Research Site, Saint-Laurent-d'Aigouze
  - Research Site, Saint-Laurent-de-la-Salanque
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Saint-Laurent-en-Grandvaux
  - Research Site, Saint-Léger-sous-Cholet
  - Research Site, Saint-Léonard-de-Noblat
  - Research Site, Saint-Loubès
  - Research Site, Saint-Marcel
  - Research Site, Saint-Marcel-lès-Valence
  - Research Site, Saint-Marcellin
  - Research Site, Saint-Martin-de-Landelles
  - Research Site, Saint-Martin-de-Valgalgues
  - Research Site, Saint-Martin-des-Champs
  - Research Site, Saint-Martin-du-Manoir
  - Research Site, Saint-Martin-du-Var
  - Research Site, Saint-Martin-en-Bresse
  - Research Site, Saint-Maur-des-Fossés
  - Research Site, Saint-Maurice-en-Gourgois
  - Research Site, Saint-Maurice-l'Exil
  - Research Site, Saint-Maurice-lès-Châteauneuf
  - Research Site, Saint-Maurice-sur-Fessard
  - Research Site, Saint-Médard-de-Guizières
  - Research Site, Saint-Michel-Chef-Chef
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Nicolas-de-Port
  - Research Site, Saint-Omer
  - Research Site, Saint-Orens-de-Gameville
  - Research Site, Saint-Ouen
  - Research Site, Saint-Pair-sur-Mer
  - Research Site, Saint-Paul-en-Chablais
  - Research Site, Saint-Paul-lès-Dax
  - Research Site, Saint-Père-en-Retz
  - Research Site, Saint-Pierre-d'Irube
  - Research Site, Saint-Pierre-des-Corps
  - Research Site, Saint-Pierre-en-Val
  - Research Site, Saint-Pierre-lès-Elbeuf
  - Research Site, Saint-Pierre-Montlimart
  - Research Site, Saint-Priest-Taurion
  - Research Site, Saint-Puy
  - Research Site, Saint-Quay-Portrieux
  - Research Site, Saint-Quentin
  - Research Site, Saint-Quentin-la-Poterie
  - Research Site, Saint-Raphaël
  - Research Site, Saint-Renan
  - Research Site, Saint-Rémy-de-Provence
  - Research Site, Saint-Romain-sur-Cher
  - Research Site, Saint-Rome-de-Cernon
  - Research Site, Saint-Sauveur
  - Research Site, Saint-Sauveur-dAunis
  - Research Site, Saint-Siméon-de-Bressieux
  - Research Site, Saint-Symphorien-sur-Coise
  - Research Site, Saint-Thégonnec
  - Research Site, Saint-Trivier-sur-Moignans
  - Research Site, Saint-Vallier
  - Research Site, Saint-Victoret
  - Research Site, Saint-Vincent-de-Mercuze
  - Research Site, Saintes
  - Research Site, Saintes-Maries-de-la-Mer
  - Research Site, Salbris
  - Research Site, Salernes
  - Research Site, Salies-de-Béarn
  - Research Site, Salies-du-Salat
  - Research Site, Salins-les-Bains
  - Research Site, Salles
  - Research Site, Salomé
  - Research Site, Salon-de-Provence
  - Research Site, Salornay-sur-Guye
  - Research Site, Sanary-sur-Mer
  - Research Site, Sarlat-la-Canéda
  - Research Site, Sarrebourg
  - Research Site, Sarreguemines
  - Research Site, Sars-Poteries
  - Research Site, Saulces-Monclin
  - Research Site, Sault
  - Research Site, Sault-lès-Rethel
  - Research Site, Sauveterre-de-Guyenne
  - Research Site, Savigny-sur-Orge
  - Research Site, Schoelcher
  - Research Site, Secondigny
  - Research Site, Sedan
  - Research Site, Seine-Port
  - Research Site, Seloncourt
  - Research Site, Seltz
  - Research Site, Semblançay
  - Research Site, Senlis
  - Research Site, Sennecey-le-Grand
  - Research Site, Sens
  - Research Site, Septfonds
  - Research Site, Seraincourt
  - Research Site, Sermoise-sur-Loire
  - Research Site, Seyssel
  - Research Site, Seyssinet-Pariset
  - Research Site, Sète
  - Research Site, Sèvres
  - Research Site, Sèvres-Anxaumont
  - Research Site, Sébazac-Concourès
  - Research Site, Sémalens
  - Research Site, Séné
  - Research Site, Sérifontaine
  - Research Site, Sigean
  - Research Site, Signy-le-Petit
  - Research Site, Simiane-Collongue
  - Research Site, Sisteron
  - Research Site, Six-Fours-les-Plages
  - Research Site, Sixt-sur-Aff
  - Research Site, Sochaux
  - Research Site, Soisy-sous-Montmorency
  - Research Site, Solliès-Toucas
  - Research Site, Solre-le-Château
  - Research Site, Songeons
  - Research Site, Sotteville-lès-Rouen
  - Research Site, Soudan
  - Research Site, Soultz-Haut-Rhin
  - Research Site, Soumoulou
  - Research Site, St-Malo
  - Research Site, St.-Jean
  - Research Site, Stains
  - Research Site, STE Fereole
  - Research Site, STE Genevieve
  - Research Site, STE Hermine
  - Research Site, STE LUCE SUR Loire
  - Research Site, STE Marie
  - Research Site, STE Maure de Touraine
  - Research Site, STE Menehould
  - Research Site, STE MERE Eglise
  - Research Site, STE Savine
  - Research Site, STE Suzanne
  - Research Site, STE Terre
  - Research Site, Strasbourg
  - Research Site, Sucy-en-Brie
  - Research Site, Tain-l'Hermitage
  - Research Site, Talange
  - Research Site, Tarare
  - Research Site, Tarbes
  - Research Site, Tardets
  - Research Site, Targon
  - Research Site, Teloché
  - Research Site, Templeuve-en-Pévèle
  - Research Site, Tencin
  - Research Site, Tergnier
  - Research Site, Teyran
  - Research Site, Thann
  - Research Site, Théoule-sur-Mer
  - Research Site, Thérouanne
  - Research Site, Thiers
  - Research Site, Thilouze
  - Research Site, Thionville
  - Research Site, Thoissey
  - Research Site, Thomery
  - Research Site, Thorigné-sur-Dué
  - Research Site, Thouarcé
  - Research Site, Thourotte
  - Research Site, Thueyts
  - Research Site, Thun-Saint-Amand
  - Research Site, Thury-Harcourt
  - Research Site, Thyez
  - Research Site, Tincques
  - Research Site, Tinqueux
  - Research Site, Toul
  - Research Site, Toulon
  - Research Site, Toulouges
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tournon-d'Agenais
  - Research Site, Tours
  - Research Site, Tourtour
  - Research Site, Trans-en-Provence
  - Research Site, Trets
  - Research Site, Trèbes
  - Research Site, Trélazé
  - Research Site, Trévoux
  - Research Site, Trith-Saint-Léger
  - Research Site, Troisfontaines
  - Research Site, Tullins
  - Research Site, Uriménil
  - Research Site, Ussel
  - Research Site, Ustaritz
  - Research Site, Uzès
  - Research Site, Vaison-la-Romaine
  - Research Site, Val-de-Saâne
  - Research Site, Valdoie
  - Research Site, Valence
  - Research Site, Valenciennes
  - Research Site, Valenton
  - Research Site, Vallauris
  - Research Site, Vallet
  - Research Site, Vallon-Pont-d'Arc
  - Research Site, Valmont
  - Research Site, Valras-Plage
  - Research Site, Valréas
  - Research Site, Vannes
  - Research Site, Varennes-Vauzelles
  - Research Site, Varreddes
  - Research Site, Vaugneray
  - Research Site, Veauche
  - Research Site, Vendenheim
  - Research Site, Vendeuil
  - Research Site, Venelles
  - Research Site, Verfeil
  - Research Site, Verneuil-en-Halatte
  - Research Site, Versailles
  - Research Site, Vesseaux
  - Research Site, Veynes
  - Research Site, Vénissieux
  - Research Site, Véretz
  - Research Site, Vézelise
  - Research Site, Vierzon
  - Research Site, Vieugy
  - Research Site, Vigneux-de-Bretagne
  - Research Site, Vigneux-sur-Seine
  - Research Site, Villeblevin
  - Research Site, Villecomtal
  - Research Site, Villedieu-les-Poêles
  - Research Site, Villefranche-sur-Saône
  - Research Site, Villemur-sur-Tarn
  - Research Site, Villeneuve les beziers
  - Research Site, Villeneuve-d'Ascq
  - Research Site, Villeneuve-la-Garenne
  - Research Site, Villeneuve-Loubet
  - Research Site, Villeneuve-Saint-Georges
  - Research Site, Villennes-sur-Seine
  - Research Site, Villepreux
  - Research Site, Villereversure
  - Research Site, Villers-Bretonneux
  - Research Site, Villers-Cotterêts
  - Research Site, Villers-Outréaux
  - Research Site, Villersexel
  - Research Site, Villeurbanne
  - Research Site, Villiers-le-Bel
  - Research Site, Villiers-Saint-Fréderic
  - Research Site, Vinay
  - Research Site, Vincennes
  - Research Site, Vinsobres
  - Research Site, Violaines
  - Research Site, Viry-Châtillon
  - Research Site, Vitrey-sur-Mance
  - Research Site, Vitrolles
  - Research Site, Vitry-en-Artois
  - Research Site, Vitry-sur-Seine
  - Research Site, Vittel
  - Research Site, Vivier-au-Court
  - Research Site, Vivy
  - Research Site, Voisins-le-Bretonneux
  - Research Site, Volgelsheim
  - Research Site, Volvic
  - Research Site, Vouneuil-sous-Biard
  - Research Site, Vouziers
  - Research Site, Vrigne-aux-Bois
  - Research Site, Vue
  - Research Site, Wailly
  - Research Site, Wallon-Cappel
  - Research Site, Wanquetin
  - Research Site, Wattignies
  - Research Site, Wattrelos
  - Research Site, Westhoffen
  - Research Site, Wignehies
  - Research Site, Wittelsheim
  - Research Site, Wittring
  - Research Site, Wolfisheim
  - Research Site, Yerres
  - Research Site, Yerville
  - Research Site, Yvetot
  - Research Site, Zillisheim
  - Research Site, Zuydcoote